CLINICAL TRIAL: NCT03816007
Title: An Enhanced Mind-body Intervention to Reduce Disability and Pain in Veterans With PTSD
Brief Title: Yoga and Mantram for Chronic Pain and PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D3009-P
Record Dates: First submitted 2019-01-17; First posted 2019-01-25 (Actual); Results first posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Post-Traumatic Stress Disorder; Chronic Low Back Pain; Chronic Neck Pain
Keywords: PTSD; chronic pain; yoga; mantram repetition; mind-body interventions; complementary and integrative medicine
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Chronic Pain | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomized to either the enhanced yoga interventions or the (R/HE) comparison intervention. Assessments will occur at baseline, 12-weeks, and again 6-weeks after the intervention ends (18-weeks). The enhanced yoga intervention will consist of 1x weekly instructor-led yoga sessions lasting approximately 75 minutes, augmented by home practice of yoga for 20 minutes/day. The R/HE control intervention will be manualized and will meet weekly for 12 weeks for approximately 75 minutes per week. Short homework assignments will be included.
Who Masked: Participant
Masking Description: Participants are blinded to which intervention is hypothesized to be superior, but are aware of the intervention they are assigned to. All assessments are self-report and do not require interpretation by study investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Yoga and Mantram Repetition (Experimental): An existing yoga intervention designed for persons with chronic pain will be augmented with training in mantram repetition. The intervention meets 1x weekly for 75 minutes for 12 weeks, and includes a home practice component.
  Interventions: Behavioral: Yoga and Mantram Repetition
- Relaxation/Health Education (Active Comparator): A relaxation intervention used previously as a comparator intervention will be delivered by a health educator.
  Interventions: Behavioral: Veteran Calm

INTERVENTIONS:
Behavioral: Yoga and Mantram Repetition — An existing yoga intervention designed for persons with chronic pain will be augmented with training in mantram repetition. The intervention meets 1x weekly for 75 minutes for 12 weeks, and includes a home practice component.
  Other Names: Yoga _+ MR
  Arms: Yoga and Mantram Repetition
Behavioral: Veteran Calm — A relaxation intervention used previously as a comparator intervention will be delivered by a health educator 1x weekly for 75 minutes for 12 weeks, and includes a home practice component.
  Other Names: VC
  Arms: Relaxation/Health Education

SUMMARY:
PTSD is prevalent among Veterans and is associated with physical and functional impairments in addition to PTSD symptoms. Veterans with PTSD experience more chronic pain and pain-related functional limitations than Veterans without PTSD. Mind-body interventions such as yoga and meditation are non-pharmacological options for treating both chronic pain and PTSD. This pilot study will add an existing mantram repetition (MR) component designed for Veterans with PTSD to an active yoga intervention known to improve function in chronic back pain patients. The study will examine the acceptability of the interventions, adverse events, and the feasibility of recruitment, attendance, retention, treatment fidelity, and assessments by recruiting and randomizing 32 VA patients with PTSD to either yoga plus MR or to a relaxation/health education control. Health outcomes including pain-related function, pain, and PTSD symptoms will be measured. If feasible, the data will be used to plan a full-scale trial of enhanced yoga for pain in VA patients with PTSD.

DETAILED DESCRIPTION:
The objectives of the proposed project are to examine the feasibility of delivering a combined yoga and MR intervention to VA patients with PTSD and cLBP and/or cNP within a randomized controlled trial study design. MR enhances the active yoga intervention for this specific population by providing a portable tool for managing stress and anxiety, and improving mental and emotional functioning in situations of daily life. The investigators will recruit and randomize 32 Veterans with PTSD to either enhanced yoga interventions or a relaxation/health education (R/HE) comparison intervention. The goal of the pilot randomized trial is to demonstrate the acceptability of the interventions, to study the feasibility of recruitment, retention, adherence, randomization, and assessments with military Veterans with PTSD, and to measure any adverse events. Data will inform plans for a full-scale effectiveness RCT.

Researchers and content experts will adapt and blend two manualized interventions (MR and yoga) into a single manualized and acceptable intervention. In addition, the existing yoga intervention and MR manuals will be adapted to provide a structured intervention guide for instructors. Next, the investigators will recruit and screen 32 Veterans with PTSD. Eligible participants will be randomized to either the enhanced yoga interventions or the (R/HE) comparison intervention. Assessments will occur at baseline, 12-weeks, and again 6-weeks after the intervention ends (18-weeks). The enhanced yoga intervention will consist of 1x weekly instructor-led yoga sessions lasting approximately 75 minutes, augmented by home practice of yoga for 20 minutes/day. The R/HE control intervention will be manualized and will meet weekly for 12 weeks for approximately 75 minutes per week. Short homework assignments will be included. The investigators will track and measure adverse events, recruitment rates, attendance and home practice rates, use of MR and yoga principles in daily life, attrition rates, and time to complete assessments. Questionnaires will assess pain-related function, pain, PTSD symptoms, insomnia/sleep, alcohol use, and quality of life. The investigators will also conduct qualitative interviews with 12 study participants to examine acceptability, recommendations, and factors affecting attendance and attrition. The investigators will target 7-8 yoga participants and 4-5 control participants. Data will be used to plan a full-scale RCT powered to detect differences in health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Veterans Affairs (VA) patients
* age > 18
* current diagnosis of PTSD
* score of 25 on Montreal Cognitive Assessment (MoCA)
* willing to reduce or cease opioid medications
* willing to attend 12-weeks of mind-body interventions and complete 3 assessments

Exclusion Criteria:

* serious or unstable psychiatric illness

  * e.g. psychosis, mania
* suicidal or homicidal ideation
* < 3 months since major trauma event
* moderate or severe cognitive impairment
* practiced yoga or mantram repetition > 2x in the last 6 months
* coexisting medical illness with yoga contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik J. Groessl, PhD BA BS, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be created and shared. Requests for access to this data must be made in writing signed by a requestor from the United States. The request should reference the publication underlying the request. Requests may be made to the Principal Investigator/lead point-of-contact for the publication. Should the investigator leave the VASDHS the requests may be sent to the VA San Diego Associate Chief of Staff for Research.
  One or more data sets without personal identifiers will be generated during the data analysis phase of this study. The data sets will include all data underlying any publications generated by this study and therefore sufficient to reproduce or verify any published findings. Publications will specify the statistical analytic methods used, thereby enabling recipients to analyze the same data and validate study results.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available within 12 months of the end of the study.
Access Criteria: Requests for access to this data must be made in writing signed by a requestor from the United States. The request should reference the publication underlying the request. Requests may be made to the Principal Investigator/lead point-of-contact for the publication. Should the investigator leave the VASDHS the requests may be sent to the VA San Diego Associate Chief of Staff for Research.

RESULTS

PARTICIPANT FLOW:
Period: End of 12-week Intervention
Arm/Group | Yoga and Mantram Repetition | Relaxation/Health Education
Started | 16 | 16
Completed | 13 | 10
Not Completed | 3 | 6
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 3 | 4
Period: Final Assessment at 18 Weeks.
Arm/Group | Yoga and Mantram Repetition | Relaxation/Health Education
Started | 16 | 14
Completed | 12 | 10
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Yoga and Mantram Repetition | Relaxation/Health Education | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (14.6) | 39.6 (10.4) | 47.1 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 4
  Male | 16 | 12 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 2 | 2 | 4
  White | 9 | 6 | 15
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Roland-Morris Disability Questionnaire (RMDQ)
Description: The RMDQ has 23 questions asking about limitations experienced with daily activities. The scale is reliable and well validated. It has been used in other yoga studies. Scores can range from 0-24. Higher scores indicate more impairment, and when considering the change from baseline to follow-up assessments, negative scores indicate improvement. The scale has been shown to be reliable and is well validated. It has been used in another yoga RCT, allowing for comparisons.
Time Frame: Change between baseline and 12-weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Yoga and Mantram Repetition | Relaxation/Health Education
Number analyzed (Participants) | 13 | 10
score on a scale | 13.6 (4.4) | 14.3 (6.6)

2. Secondary Outcome: BPI Pain Severity
Description: Brief Pain Inventory Pain Severity - The total score is the mean of the 4 pain severity items. Scores range from 0-10 with higher scores indicating greater pain severity.
Time Frame: change from baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Yoga and Mantram Repetition | Relaxation/Health Education
Number analyzed (Participants) | 13 | 10
score on a scale | -0.15 (1.71) | -1.15 (1.78)

3. Secondary Outcome: Post-Traumatic Stress Disorder Checklist- Version 5 (PCL-5)
Description: The PCL-5 is a 20-item self-report measure assessing 20 DSM-5 symptoms of PTSD. Each question is rated on a scale from 0-4 and the total score ranges from 0-80 with higher scores indicating a greater severity of PTSD symptoms.
Time Frame: Change between baseline and 12-weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Yoga and Mantram Repetition | Relaxation/Health Education
Number analyzed (Participants) | 13 | 10
score on a scale | -4.23 (13.8) | -9.80 (12.6)

4. Secondary Outcome: BPI Pain Interference
Description: Brief Pain Inventory Pain Interference - The total score is the mean of the 7 pain interference items. Scores range from 0-10 with higher scores indicating greater pain interference.
Time Frame: change from baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Yoga and Mantram Repetition | Relaxation/Health Education
Number analyzed (Participants) | 13 | 10
score on a scale | -0.73 (2.28) | -0.46 (2.24)

5. Secondary Outcome: Insomnia Severity Index (ISI)
Description: Insomnia Severity Index is a 7-item instrument that assesses the impact of insomnia. Each question is rated on a scale from 0-4 and the total score ranges from 0-28 with higher scores indicating a greater severity of insomnia.
Time Frame: Change between baseline and 12-weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Yoga and Mantram Repetition | Relaxation/Health Education
Number analyzed (Participants) | 13 | 10
score on a scale | -2.69 (7.18) | -0.30 (3.92)

6. Secondary Outcome: Quality of Life - EQ5D
Description: Health-related Quality of Life will be measured with the EQ5D-3L. Scores range from 0 to 1.0 with higher scores indicating better quality of life.
Time Frame: Change between baseline and 12-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yoga and Mantram Repetition | Relaxation/Health Education
Number analyzed (Participants) | 13 | 10
units on a scale | 0.02 (0.22) | 0.10 (0.28)

7. Secondary Outcome: AUDIT-C
Description: AUDIT-C is a 3-item screen for problem drinking and will refer to alcohol use over the past 3-month period. The measure has questions on typical consumption and binge drinking frequency. Each question is rated on a scale from 0-4 and the total score ranges from 0-12 with higher scores indicating a greater likelihood of alcohol use problems.
Time Frame: Change between baseline and 12-weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Yoga and Mantram Repetition | Relaxation/Health Education
Number analyzed (Participants) | 13 | 10
score on a scale | -0.62 (0.87) | -0.10 (0.57)

8. Secondary Outcome: Fatigue
Description: Fatigue Severity Scale - The scale consists of 9 items describing the functional impact of fatigue on daily life rated on a scale from 1 (strongly disagree) to 7 (strongly agree) with the total fatigue score ranging from 9-63. Higher scores reflect greater fatigue severity and less energy.
Time Frame: change from baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Yoga and Mantram Repetition | Relaxation/Health Education
Number analyzed (Participants) | 13 | 10
score on a scale | -7.38 (9.38) | -4.90 (8.16)

ADVERSE EVENTS:
Time Frame: from baseline to 18-week follow-up assessment
Arm/Group | Yoga and Mantram Repetition | Relaxation/Health Education
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 3/16 | 0/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Yoga and Mantram Repetition (N=16) | Relaxation/Health Education (N=16)
muscle and joint soreness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
recurring back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ongoing numbness and tingling in arm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/07/NCT03816007/Prot_SAP_001.pdf
  • Informed Consent Form (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/07/NCT03816007/ICF_000.pdf